CLINICAL TRIAL: NCT03996772
Title: PREvention of STroke in Intracerebral haemorrhaGE Survivors With Atrial Fibrillation (PRESTIGE-AF)
Brief Title: PREvention of STroke in Intracerebral haemorrhaGE Survivors With Atrial Fibrillation
Acronym: PRESTIGE-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Wuerzburg University Hospital (Other); Julius-Maximilians University (Other); Medical University of Graz (Other); University of Liverpool (Other); King's College London (Other); Hospital Universitari Vall d'Hebron Research Institute (Other); University of Bordeaux (Other); Azienda Ospedaliera di Perugia (Other); Aalborg University (Other); STROKE ALLIANCE FOR EUROPE (Unknown); University Hospital Heidelberg (Other); Imperial College Healthcare NHS Trust (Other); Alfried Krupp Krankenhaus (Other); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17HH4268; 2018-002176-41 (EudraCT Number); 754517 (Other Grant/Funding Number: European Union Horizon 2020); 236886 (Other: IRAS)
Record Dates: First submitted 2019-06-03; First posted 2019-06-25 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Atrial Fibrillation; Intracerebral Hemorrhage
Keywords: Atrial fibrillation; Arrhythmias; Cardiac; Cerebral Hemorrhage; Brain haemorrhage; Intracerebral hemorrhage; Cerebral haemorrhage; Basal ganglia haemorrhage; Putaminal haemorrhage; Anticoagulants; Oral anticoagulant; Direct oral anticoagulant; New oral anticoagulant; Factor Xa inhibitors; Direct thrombin inhibitor; Dabigatran; Apixaban; Rivaroxaban; Edoxaban; DOAC; NOAC; Intracerebral haemorrhage; Brain hemorrhage
MeSH Terms: conditions — Atrial Fibrillation; Cerebral Hemorrhage; Arrhythmias, Cardiac; Intracranial Hemorrhages; Basal Ganglia Hemorrhage | interventions — apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: PREvention of STroke in Intracerebral haemorrhaGE survivors with Atrial Fibrillation is a phase 3b investigator-led, multicentre, parallel group, prospective randomised, open, blinded end-point assessment (PROBE) clinical trial comparing direct oral anticoagulants against no anticoagulation in patients with a recent intracerebral haemorrhage (ICH) and comorbid atrial fibrillation (AF).
  Randomisation will occur in a 1:1 ratio. Participants will be stratified according to two factors: lobar and non-lobar location of ICH and gender. Choice and dose of direct oral anticoagulant treatment and use of concomitant medication during the study treatment will be at the Principal Investigator´s discretion within the licensed doses for stroke prevention in AF patients in Europe. The control group will receive no anticoagulant but the use of an antiplatelet is at the Principal Investigator´s discretion who will use their clinical judgment to initiate an antiplatelet drug of their choice.
Who Masked: Outcomes Assessor
Masking Description: An Event Adjudication Committee (EAC) will be established. The EAC will consist of experts in relevant fields of the Study such as neurology, cardiology, and haematology. An event adjudication charter with clear definitions of pre-specified outcome events will be developed by the steering committee and agreed by the EAC. After formal training, the EAC will be provided with pseudonymised data for adjudication of pre-specified outcome events and serious adverse events using an online platform provided by the data management centre, Clinical Trials Center Wuerzburg at the University of Wuerzburg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Direct Oral Anticoagulant (Experimental): If the patient is randomized in this arm, a direct oral anticoagulant (DOAC) included:
  * Direct thrombin inhibitor: Dabigatran
  * Factor Xa inhibitors: Apixaban or Rivaroxaban or Edoxaban will be prescribed to the patient. Choice and dose of DOAC treatment as well as the use of concomitant medication during the study treatment will be at the Principal Investigator´s discretion within the spectrum of licensed doses labelled for stroke prevention in atrial fibrillation patients in Europe following the Summary of Product Characteristics.
  Interventions: Drug: Apixaban Oral Tablet; Drug: Dabigatran; Drug: Edoxaban Tablets; Drug: Rivaroxaban
- No Anticoagulant (No Intervention): If the patient is randomized in this arm investigators will use their best judgment to decide upon the prescription of an antiplatelet drug of their choice or no such therapy

INTERVENTIONS:
Drug: Apixaban Oral Tablet — Factor Xa Inhibitor
  Other Names: Eliquis
  Arms: Direct Oral Anticoagulant
Drug: Dabigatran — Direct Thrombin Inhibitor
  Other Names: Pradaxa
  Arms: Direct Oral Anticoagulant
Drug: Edoxaban Tablets — Factor Xa Inhibitor
  Other Names: Lixiana; Savaysa
  Arms: Direct Oral Anticoagulant
Drug: Rivaroxaban — Factor Xa Inhibitor
  Other Names: Xarelto
  Arms: Direct Oral Anticoagulant

SUMMARY:
Atrial fibrillation (AF) is the most common form of irregular heart rhythm. In people with AF, blood clots often form in the heart, which can travel to the brain. Blockage of brain arteries by these clots is a major cause of stroke. This type of stroke is called an ischaemic stroke and approximately 15% of all ischaemic strokes are caused by AF.

People with AF are often prescribed a medication called an anticoagulant, which makes it less likely for blood clots to form and thus can prevent ischaemic strokes. However, anticoagulants also increase the risk of bleeding, so they are not suitable for everyone.

Some people who have AF have had a different type of stroke which is caused by bleeding in the brain, an intracerebral haemorrhage (ICH). These people are at increased risk of suffering both an ischaemic stroke (due to AF) and another ICH. It is not known whether it is best for these people to take an anticoagulant medication or not, as previous research studies did not include this group of people.

PREvention of STroke in Intracerebral haemorrhaGE survivors with Atrial Fibrillation (PRESTIGE-AF) is a research study on the best stroke prevention in people with atrial fibrillation (AF) who have recently had a bleeding in their brain, (ICH). This is a trial where half of the participants will take an anticoagulant medication, preventing blood clot formation, and half will not receive an anticoagulant. The direct oral anticoagulants (DOACs) that will be used in this trial are all licenced for use in the United Kingdom and within the European Union (EU) to prevent strokes in people with AF. However, the current licence does not extend to use with people who have had an ICH because it has not been tested in this group with a randomised controlled trial. DOACs will be tested in ICH survivors with AF because previous research trials have shown that people are up to 50% less likely to have bleeding complications in the brain with DOACs than with Warfarin (another commonly used anticoagulant).

The aim of PRESTIGE-AF is to answer the question of whether people with ICH and AF should take an anticoagulant medication or if it is better for them to avoid it.

DETAILED DESCRIPTION:
Stroke is one of the largest public health challenges worldwide. Its societal impact is expected to further increase in the coming decades due to the aging of population. Importantly, stroke is a heterogeneous disease comprising various subtypes with distinct mechanisms. The variability of individual risks demands that more specifically targeted and better personalised approaches are developed to tailor stroke prevention for particular stroke types and individual patients.

Intracerebral haemorrhage (ICH) is a particularly severe type of stroke affecting 10-15% of all stroke patients. Importantly, ICH carries even higher mortality and more severe disability than other stroke types. While mechanisms of ICH and ischaemic stroke are distinct, many risk factors are shared and patients are often at increased risk of both ischaemic stroke and ICH.

Atrial fibrillation (AF) is also a growing epidemic in aging populations and a major cause of ischaemic stroke due to thrombus formation in the heart migrating to and occluding intracerebral arteries. At least 20% of ICH survivors also suffer from AF and are, thus, at particularly high risk of ischaemic stroke. While ischaemic stroke in AF patients in general can be much more effectively prevented with oral anticoagulation than with antiplatelet agents (APA) concerns about ICH recurrence in ICH survivors are a major barrier for anticoagulation. The best approach to stroke prevention in ICH patients with AF is presently unknown. Current clinical guidelines, which are largely based on retrospective observational studies investigating anticoagulation with vitamin K antagonists (VKA), either recommend considering anticoagulation only in patients with non-lobar location of ICH or, in the absence of evidence from randomised controlled trials, refrain from making any recommendations at all. Anticoagulation with direct oral anticoagulants (DOAC) has proven efficacy and safety for stroke prevention in AF. DOACs may be a better alternative to VKA particularly in ICH patients because DOACs were associated with a 50% lower risk of ICH than VKA in previous clinical trials of stroke prevention in AF. However, patients with previous ICH were excluded from these trials.

Although thousands of ICH survivors with AF every year worldwide need effective prevention of another stroke, the best antithrombotic therapy for these patients is currently unknown. PRESTIGE-AF will be the first sufficiently powered randomised controlled trial aiming to resolve the dilemma of stroke prevention in this challenging high-risk patient population. Specifically, it will answer the question whether DOAC with their well-documented lower risk of intracranial haemorrhagic complications, compared to VKA, provide both a more effective and an equally safe option for stroke prevention in patients with ICH and AF compared to no anticoagulant. Findings of the Study are expected to change management guidelines and future prevention research for ICH survivors with AF.

PREvention of STroke in Intracerebral haemorrhaGE survivors (PRESTIGE-AF) will test whether preventive therapy with DOACs (intervention group) reduce the rate of ischaemic stroke (superiority) compared to no anticoagulation (control group) without unacceptably increasing the risk of recurrent ICH (non-inferiority) in patients with AF and a previous ICH within 6 months before enrolment.

The Research Question is:

Does preventive therapy with Direct Oral Anticoagulants (intervention group) reduce the rate of ischaemic stroke (superiority) compared to no anticoagulation (control group) without unacceptably increasing the risk of recurrent Intracerebral haemorrhage (non-inferiority) in patients with atrial fibrillation and a previous intracerebral haemorrhage within 6 months before enrolment.

The Objectives of the study are:

The main objective is to perform a randomised controlled trial to resolve the long-standing management dilemma of antithrombotic stroke prevention in intracerebral haemorrhage (ICH) survivors with comorbid atrial fibrillation (AF). Specifically, it will address the question whether direct oral anticoagulants (DOACs, intervention) provide a more effective option for prevention of ischaemic stroke and an equally safe option in terms of recurrence of ICH for antithrombotic stroke prevention in survivors of recent ICH compared to no anticoagulation (i.e. no antithrombotic therapy or antiplatelet therapy at Principal Investigator´s discretion).

The secondary Study objectives are:

* To examine the effect of anticoagulation with DOAC versus no anticoagulation on major cardiovascular outcomes and mortality in ICH patient with AF
* To compare the effect of DOACs versus no anticoagulation on major systemic and intracranial bleeding in this Study population
* To examine the effect of DOACs versus no anticoagulation on net clinical benefit in ICH patients with AF

The exploratory objectives are:

• To explore the impact of DOAC vs. no anticoagulation on quality of life, cognition and psychological morbidity in patients with ICH and AF over time Study Design: PRESTIGE-AF is a phase 3b investigator-led, multicentre, parallel group, prospective randomised, open, blinded end-point assessment (PROBE) clinical trial comparing DOACs (interventional arm) against no anticoagulation (control arm) in patients with a recent ICH and comorbid AF.

Randomisation will occur in a 1:1 ratio. Participants will be stratified according to two factors: lobar and non-lobar location of ICH and sex. Choice and dose of DOAC treatment as well as the use of concomitant medication during the study treatment will be at the Principal Investigator´s discretion within the spectrum of licensed doses labelled for stroke prevention in AF patients in Europe following the Summary of Product Characteristics (SmPC). The control group will receive no anticoagulant but the use of an antiplatelet agent is at the Principal Investigator´s discretion who will use their clinical judgment to initiate (or not) an antiplatelet drug of their choice.

Baseline assessment will include capturing Participant's demographics, clinical characteristics, vital signs, medical history, and concomitant diseases as well as documentation of AF (previous history or newly detected). Results of routine diagnostic tests before Study enrolment will be also collected using an electronic case report form. The routine brain imaging data performed after the ICH and before Study enrolment will also be collected at baseline.

After randomisation, Participants will be followed-up in person at various time points (1, 6, 12, 24, 36 months) for up to 3 years. At each visit, outcome events and adverse events will be captured.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent obtained from the patient, or for patients who lack the capacity to consent this can be provided by an appropriate representative as defined in protocol
* Non-traumatic spontaneous ICH during the 12 months before enrolment. Patients become eligible 14 days after the date of their ICH.
* Documented evidence of AF (paroxysmal, persistent or permanent)

Exclusion Criteria:

* Fully dependent (mRS >4)
* Women who are pregnant, breastfeeding, or plan to become pregnant during the Study period
* Women of childbearing potential (WOCBP see section 12.2 for definition) who are unable or unwilling to take measures for effective contraception (4.9)
* Enrolment occurring before 14 days after the date of ICH
* Enrolment occurring longer than 12 months after the date of ICH
* ICH resulting from trauma or vascular malformation
* Another indication for long-term anticoagulation
* Patient has hypertension, which in the opinion of the investigator, is uncontrollable with medication Any contraindication (except intracerebral haemorrhage) to treatment with apixaban, dabigatran, edoxaban, rivaroxaban as per SmPC. Including any of the following:

  * Hypersensitivity to the active principle or any of the excipients
  * Clinically relevant bleeding in progress
  * Liver disease associated with coagulopathy and a clinically relevant bleeding risk
  * Injuries or conditions such as a significant risk of major bleeding
  * Hepatic impairment or liver disease which can have an impact on survival
  * Exclusion of patients with end-stage renal creatinine clearance CrCL, (CrCL <15 ml / min) or in patients undergoing dialysis
  * Concomitant treatment with other anticoagulants
  * Patients with a history of thrombosis and antiphospholipid antibody syndrome Special warnings and precautions for use for apixaban, dabigatran, edoxaban, rivaroxaban as per SmPC should also be taken into account at randomisation.
* Absolute need for antiplatelet agent (APA) at enrolment, meaning that a patient randomised to receive DOAC who would require an APA is not eligible (single APA is permitted in control group only, at time of randomisation). Presence of a left atrial appendage occlusion device (LAAO) or plan to implant an LAAO
* Presence of any medical, psychological, or psychiatric condition which in the opinion of the Principal or Co-Investigator would cause participation in the Study to be unwise
* Participation in any clinical study with an Investigational Medicinal Product within the past 30 days or 5 half-lives of the study drug (observational studies are permitted)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Time to the first incident ischemic stroke event. | 3 years
  Statistics: product-limit estimations of the time to event ("survival") functions in both study groups. Measure of association: hazard ratio under the proportional hazard assumption.
Time to the first recurrent intracerebral haemorrhage event. | 3 years
  Statistics: product-limit estimations of the time to event ("survival") functions in both study groups. Measure of association: hazard ratio under the proportional hazard assumption.

SECONDARY OUTCOMES:
Rate of all stroke events | 3 years
  Rate of all stroke events from the index date as number of events per 100 person years under observation in the study
Rate of systemic embolism | 3 years
  Rate of systemic embolism from the index date as number of events per 100 person years under observation in the study
Rate of major adverse cardiac events | 3 years
  Rate of major adverse cardiac events from the index date as number of events per 100 person years under observation in the study
Rate of all-cause mortality | 3 years
  Rate of all-cause mortality from the index date as number of events per 100 person years under observation in the study
Rate of cardiovascular mortality | 3 years
  Rate of cardiovascular mortality from the index date as number of events per 100 person years under observation in the study
Rate of major haemorrhage | 3 years
  Rate of major haemorrhage from the index date as number of events per 100 person years under observation in the study
Rate of any intracranial haemorrhage | 3 years
  Rate of any intracranial haemorrhage from the index date as number of events per 100 person years under observation in the study
Rates of events (all strokes, systemic embolic event, myocardial infarction, cardiovascular mortality and major bleeding) | 3 years
  Rates of events (all strokes, systemic embolic event, myocardial infarction, cardiovascular mortality and major bleeding) from the index date as number of events per 100 person years under observation in the study
Rate of myocardial infarction | 3 years
  Rate of myocardial infarction from the index date as number of events per 100 person years under observation in the study
Rate of major bleedings | 3 years
  Rate of major bleedings from the index date as number of events per 100 person years under observation in the study
Quality of life: EQ-5D | enrolment visit, 6 months (min follow-up), 12 months, 24 months, 36 months, and End of Treatment Visit (between 6 and 36 Months).
  Quality of life: EQ-5D with 3 levels of severity for each of the 5 dimensions:
  EQ-5D-3L
  Statistics at 12, 24 (if required) and 36 months (if required) in both study groups:
  Measures of central tendency and dispersion (mean and SD resp. median and interquartile range) for EQ VAS score (range 0 -100, higher values considered to be a better outcome) and for the EQ-5D-3L index score (range 0 - 1, higher values considered to be a better outcome) health profile: numbers and proportions reporting frequencies of the three levels within the EQ-5D dimensions in both study groups
Cognitive function: the Montreal Cognitive Assessment (MoCA) | enrolment visit, 6 months (min follow-up), 12 months, 24 months, 36 months, and End of Treatment Visit (between 6 and 36 Months).
  Cognitive function: the Montreal Cognitive Assessment (MoCA) Total MoCA score: Range: 0 - 30, higher values considered to be a better outcome.
  Statistics at 12, 24 (if required) and 36 months (if required) in both study groups:
  Measures of central tendency and dispersion (mean and SD resp. median and inter quartile range). Frequencies for the values of the subscores in both study groups
Psychological morbidity: the Hospital Anxiety and Depression Scale (HADS) | enrolment visit, 6 months (min follow-up), 12 months, 24 months, 36 months, and End of Treatment Visit (between 6 and 36 months).
  Psychological morbidity: the Hospital Anxiety and Depression Scale (HADS) Statistics at 12, 24 (if required) and 36 months (if required) in both study groups.
  HADS anxiety and HADS depression score. For both scales range 0 - 21, smaller values considered to be a better outcome.
  Median score and interquartile range for both scales in both study groups. Numbers and percentages of those patients classified as "non-cases", having mild disease, having moderate disease and having severe disease for both scales in both study groups according to the cut-off scores for HADS quantification.

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Veltkamp, FESO, Principal Investigator — Imperial College London
Locations (64):
- Austria (4):
  - Krankenhaus der Barmherzigen Brüder Eisenstadt, Eisenstadt
  - Medizinische Universität Graz, Graz
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Universitätsklinikum St. Pölten, Sankt Pölten
- France (2):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Caen Normandie, Caen
- Germany (25):
  - Universitätsklinikum Aachen, Aachen
  - Klinikum Altenburger Land, Altenburg
  - Universitätsklinikum Augsburg, Augsburg
  - Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Vivantes Hospital Neukolin, Berlin
  - Universitätsklinikum Knappschaftskrankenhaus Bochum, Bochum
  - Knappschaftskrankenhaus Bottrop, Bottrop
  - University Hospital Cologne, Cologne
  - Klinikum Dortmund, Dortmund
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - University Hospital Erlangen, Erlangen
  - Alfried Krupp Von Bohlen und Halbach-Krankenhaus, Essen
  - University Hospital Frankfurt, Frankfurt
  - Universitiaetsklinikum Giessen und Marburg (UKGM) - Standort Giessen, Geißen
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Medizinische Hochschule Hannover, Hanover
  - University Hospital Heidelberg, Heidelberg
  - University of Leipzig, Leipzig
  - University Hospital Schleswig-Holstein Campus Luebeck, Lübeck
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Landeshauptstadt Stuttgart, Stuttgart
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Universitätsklinikum Wuerzburg, Würzburg
- Italy (11):
  - Azienda USL Umbria 1 - Ospedale di Branca-Gubbio, Branca
  - Ospedale Bufalini di Cesena, Cesena
  - Azienda USL Umbria 1 - Ospedale di Città di Castello, Città di Castello
  - Azienda USL Umbria 2, Foligno
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Istituto Clinico Humanitas, Milan
  - Azienda Ospedaliera di Rilievo Nazionale (A.O.R.N) A. Cardarelli di Napoli, Napoli
  - Azienda Ospedaliera di Perugia, Perugia
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera S Camillo Forlanini, Rome
  - Azienda Ospedaliera Universitaria Senese, Siena
- Spain (10):
  - Hospital Universitario Torrecárdenas, Almería
  - Fundacío Institut d'Investigacío Biomèdica de Bellvitge, Barcelona
  - Hospital Germans Trias I Pujol, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Dr Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid
  - Complejo Hospitalario Universitario de Santiago, Santiago
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (12):
  - East Kent Hospitals University NHS Foundation Trust, Ashford
  - Northumbria Healthcare NHS Foundation Trust, Ashington
  - Basildon and Thurrock University Hospitals NHS Trust, Basildon
  - Cambridge University Hospitals NHS Trust, Cambridge
  - Countess of Chester Hospital, Chester
  - Hull and East Yorkshire NHS Trust, Hull
  - Kings College Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - St Helens and Knowsley Teaching Hospital NHS Trust, Prescot
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - Mid Yorkshire Hospitals NHS Trust, Wakefield
  - West Hertfordshire Hospitals NHS Trust, Watford

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to PRESTIGE-AF collaborators who are listed in the collaborators section. This is necessary to undertake the work as stipulated in the Grant Agreement with the European Union for this Project.
Supporting Information: Study Protocol, CSR
Time Frame: The data will be available to PRESTIGE-AF collaborators from end of data collection and will be available throughout the archive period (15 years) through the archive system.
Access Criteria: According to Study Protocol

REFERENCES:
- [Derived] Fandler-Hofler S, Ropele S, Gattringer T, Haidegger M, Pinter D, Kneihsl M, Korompoki E, Montaner J, Caso V, Ringleb PA, Sibon I, Halse O, Harvey K, Fiessler C, Wolfe CDA, Heuschmann PU, Veltkamp R, Enzinger C; PRESTIGE-AF Consortium. Neuroimaging Markers Associated With Recurrent Stroke in Intracerebral Hemorrhage and Atrial Fibrillation: Secondary Analysis of PRESTIGE-AF. Neurology. 2025 Dec 9;105(11):e214386. doi: 10.1212/WNL.0000000000214386. Epub 2025 Nov 6. PMID 41197104
- [Derived] Veltkamp R, Korompoki E, Harvey KH, Harvey ER, Fiessler C, Malzahn U, Rucker V, Montaner J, Caso V, Sibon I, Ringleb P, Halse O, Hugen K, Ullmann S, Schuhmann C, Todd GP, Haas K, Pala E, Debette S, Lachaize M, D'Aoust T, Enzinger C, Ropele S, Fandler-Hofler S, Haidegger M, Wang Y, Wafa HA, Cancelloni V, Mosconi MG, Lip GYH, Lane DA, Haefeli WE, Foerster KI, Wurmbach VS, Nielsen PB, Hajjar K, Muller P, Poli S, Purrucker J, Laible M, D'Anna L, Silva Y, de Torres Chacon R, Martinez-Sanchez P, Boulanger M, Norrving B, Pare G, Wachter R, Ntaios G, Wolfe CDA, Heuschmann PU; PRESTIGE-AF Consortium. Direct oral anticoagulants versus no anticoagulation for the prevention of stroke in survivors of intracerebral haemorrhage with atrial fibrillation (PRESTIGE-AF): a multicentre, open-label, randomised, phase 3 trial. Lancet. 2025 Mar 15;405(10482):927-936. doi: 10.1016/S0140-6736(25)00333-2. Epub 2025 Feb 26. PMID 40023176
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170